CLINICAL TRIAL: NCT01665742
Title: Novel Anti-inflammatory Dietary Intervention to Improve the Metabolic Phenotype of Overweight and Obese 13-18 Year Old Adolescents - Insights Into Potential Genetic Susceptibility
Brief Title: Anti-inflammatory Dietary Intervention in Overweight and Obese Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University College Dublin (Other)
Collaborators: National Children's Research Centre, Ireland (Network); University of Dublin, Trinity College (Other); The Adelaide and Meath Hospital (Other); St. James's Hospital, Ireland (Other)
Responsible Party: Principal Investigator, Prof Helen M Roche, Associate Professor of Nutrigenomics, University College Dublin
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TNS-5
Record Dates: First submitted 2012-08-12; First posted 2012-08-15 (Estimated); Last update posted 2014-12-09 (Estimated); Status verified 2014-12

CONDITIONS: Overweight; Obesity
Keywords: Obesity; Chronic inflammation; Anti-inflammatory dietary intervention; Genetic susceptibility
MeSH Terms: conditions — Overweight; Obesity; Genetic Predisposition to Disease | interventions — Ascorbic Acid; alpha-Tocopherol; Tea; Lycopene

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Anti-inflammatory supplement (Active Comparator): 8-weeks of daily supplementation with:
  1 x fruit juice fortified with fish oil, and 4 x film-coated tablets containing vitamin C, alpha-tocopherol, green tea extract and lycopene
  in conjunction with a weight management programme
  Interventions: Dietary Supplement: Supplement containing fish oil, vitamin C, alpha-tocopherol, green tea extract and lycopene
- Placebo supplement (Placebo Comparator): 8 weeks of daily supplementation with:
  1 x fruit juice fortified with high-oleic sunflower oil, and 4 x film-coated placebo tablets
  in conjunction with a weight management programme
  Interventions: Dietary Supplement: Placebo supplement

INTERVENTIONS:
Dietary Supplement: Supplement containing fish oil, vitamin C, alpha-tocopherol, green tea extract and lycopene — 1 x fruit juice fortified with salmon oil containing 1000mg EPA and 1000mg DHA daily for 8 weeks
  AND
  4 x film-coated tablets containing 561mg vitamin C, 389mg alpha-tocopherol, 416mg green tea extract and 15mg lycopene daily for 8 weeks
  in conjunction with a weight management programme
  Arms: Anti-inflammatory supplement
Dietary Supplement: Placebo supplement — 1 x fruit juice fortified fortified with high oleic sunflower oil daily for 8 weeks
  AND
  4 x film-coated placebo tablets daily for 8 weeks
  in conjunction with a weight management programme
  Arms: Placebo supplement

SUMMARY:
The number of overweight and obese children has increased in Ireland at a greater rate than worldwide trends. The poor eating patterns that drive adolescent obesity leads to an increase in the number of unhealthy inflammatory hormones and fats circulating in the blood which increase an adolescent's risk of developing diabetes and heart disease later in life. Dietary patterns have changed whereby key nutrients that are found in fruit, vegetables and fish, which are known to have beneficial effects and reduce risk of obesity and diabetes in later life, may need to be replaced. This project will determine whether a key anti-inflammatory nutrient supplement taken for 8 weeks will improve the metabolic profile of adolescents aged 13-18 years old. Detailed cellular analysis will determine the cellular and molecular mechanisms to provide a thorough explanation of the health effects of this intervention.

DETAILED DESCRIPTION:
The emerging model of obesity and diabetes is characterised by sub-acute chronic inflammation and insulin resistance. Mechanistic data indicates inflamed adipose tissue with increased infiltration of immune cells that generate pro-inflammatory cytokines. With childhood obesity in Ireland increasing at a rapid pace, it is important to establish the role of a non-pharmacological dietary approach to decreasing the sub-acute chronic inflammation seen in overweight and obese children. Several foods contain nutrients that are known to have anti-inflammatory properties. Such foods including fish, fruits and vegetables are known to be deplete in the adolescent diet. The aim of this project is to investigate whether a nutritional supplement containing anti-inflammatory nutrients, n-3 polyunsaturated fatty acids (found in fish oil), vitamin C, vitamin E, and polyphenols found in green tea and tomato; will improve metabolic phenotype in 13-18 year old teenagers over an 8-week period. Further, to provide insight into the role of genetics in the development of metabolic dysregulation and response to dietary treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female
2. 13-18 years
3. Body mass index ≥ 91st percentile on UK growth reference charts (Cole, 1995)
4. Medications/dietary supplements which do not interfere with the intervention are allowed, on condition that the participants adhere to the same regimen during the intervention, including oral contraceptives and other non-fatty acid based dietary supplements (e.g. garlic)
5. Smoker or non-smoker
6. Not participating in any other intervention study

Exclusion Criteria:

1. Pregnancy or lactation
2. Endocrine disorders such as Polycystic Ovary Syndrome
3. Currently on treatment for a chronic inflammatory condition such as asthma
4. Kidney or liver dysfunction
5. Iron deficiency anaemia
6. Prescribed anti-inflammatory medication
7. Consumers of fatty acid supplements including fish oils, evening primrose oil and antioxidant vitamin (A, C, E, -carotene) supplements
8. High consumers of oily fish (> 2 servings/week)
9. Participants planning to start a special diet or lose weight (e.g. Slimfast, Atkins etc)
10. Weight change ≥3kg within the last 3 months
11. Alcohol or drug abuse (based on clinical judgement)
12. Participants with an allergy to fish and/or shellfish

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 58 (Actual)
Dates: Start 2012-01; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Homeostasis model of assessment - insulin resistance | 8 weeks
  Homeostasis model of assessment - insulin resistance (HOMA-IR) will be derived from fasting glucose and insulin concentrations [(fasting plasma glucose x fasting serum insulin)/22.5] as determined by Matthews et al., 1985

SECONDARY OUTCOMES:
Adiponectin | 8 weeks
  Adiponectin, a marker of insulin sensitivity, will be determined pre- and post-intervention.
Markers of inflammation | 8 weeks
  Markers of inflammation such as C reactive protein, interleukin (IL) - 6, IL-1β, tumour necrosis factor alpha, intra-cellular adhesion molecule-1, vascular cell adhesion molecule-1, retinol binding protein 4, fibrinogen, white blood cells and related inflammatory markers
Lipid Profile | 8 weeks
  Full lipid profile and lipidomic analyses (total triacylglycerol, non-esterified fatty acids, total cholesterol, LDL cholesterol, HDL cholesterol and plasma fatty acid composition, diglycerides, cholesterol esters and sphingomyelins,) and related lipid markers
Inflammatory genetic variants | 8 weeks
  Inflammatory genetic variants such as complement component 3, lymphotoxin- α, IL-6, IL-1β, TNF-α, adiponectin polymorphisms and related variants that link to the inflammatory phenotype
Functional molecular analysis (ex-vivo) | 8 weeks
  Functional molecular analysis will be conducted to determine which insulin sensitising pathways have been modulated by the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Helen M Roche, BSc, MSc, PhD, Principal Investigator — University College Dublin; Fiona Lithander, BSc, PhD, Principal Investigator — University of Dublin, Trinity College
Locations (3):
- Ireland (3):
  - Adelaide and Meath Hospital, Incorporating the National Children's Hospital Dublin,, Dublin
  - Trinity Centre for Health Sciences, St, James's Hospital, Dublin
  - University College Dublin, Dublin

REFERENCES:
- [Derived] McMorrow AM, Connaughton RM, Magalhaes TR, McGillicuddy FC, Hughes MF, Cheishvili D, Morine MJ, Ennis S, Healy ML, Roche EF, Tremblay RE, Szyf M, Lithander FE, Roche HM. Personalized Cardio-Metabolic Responses to an Anti-Inflammatory Nutrition Intervention in Obese Adolescents: A Randomized Controlled Crossover Trial. Mol Nutr Food Res. 2018 May;62(10):e1701008. doi: 10.1002/mnfr.201701008. PMID 29665620